CLINICAL TRIAL: NCT05825456
Title: Metastatic Pathologic Fractures: Short Term Results of Endoprosthetic Reconstruction, Intramedullary Nail and Open Reduction Internal Fixation
Brief Title: Metastatic Pathologic Fractures, Short Term Results
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Merve Dursun Savran, MD, MD, Ankara University
Other Study IDs: AnkaraUniOrtho
Record Dates: First submitted 2023-03-26; First posted 2023-04-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Pathologic Fracture; Bone Metastases; Metastatic Cancer
Keywords: bone metastasis; pathologic fracture; endoprosthetic reconstruction; intramedullary nailing; open reduction internal fixation; plate and screws
MeSH Terms: conditions — Fractures, Spontaneous; Neoplasm Metastasis | interventions — Fracture Fixation, Intramedullary; Bone Plates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- endoprosthetic reconstruction: This is the group of patients with metastatic pathologic fractures treated with endoprosthesis. For example, proximal femur prosthesis for femoral neck fractures.
  Interventions: Procedure: endoprosthetic reconstruction
- intramedullary nail: This is the group of patients with metastatic pathologic fractures treated with intramedullary nail, and additional bone cement if needed. For example, proximal femur nail for trochanteric fractures, or long femoral nail for femoral shaft fractures.
  Interventions: Procedure: Intramedullary nailing
- open reduction internal fixation with plate and screws: This is the group of patients with metastatic pathologic fractures treated with open reduction internal fixation; with plates and screws. For example, reconstruction plates for pelvic fractures or 3.5 locking compression plates for humeral or femur shaft fractures.
  Interventions: Procedure: Open reduction internal fixation with plate and screws

INTERVENTIONS:
Procedure: endoprosthetic reconstruction — This is a type of surgery in which the affected part of the bone and joint is removed, and replaced by a prosthesis.
  Groups: endoprosthetic reconstruction
Procedure: Intramedullary nailing — This is a type of surgery in which the affected bone is stabilized by a nail. The affected part could be removed or retained. If removed, the defect is filled with bone cement.
  Groups: intramedullary nail
Procedure: Open reduction internal fixation with plate and screws — This is a type of surgery in which the affected part of the bone is visualized completely, after the reduction is achieved, the fixation is provided with appropriate plates and screws. Again the affected part could be removed or retained. If removed, the defect is filled with bone cement.
  Groups: open reduction internal fixation with plate and screws

SUMMARY:
This is a single center prospective study to compare the short term results of prosthesis, nail and plate-screw surgeries for metastatic pathologic fractures.

DETAILED DESCRIPTION:
The most common bone tumor in elderly is metastatic bone tumors. With the prolonged life expectancy in cancer patients, the management of the metastases became an essential topic.

Pathological fractures should be examined and managed with a different perspective. They usually cannot be healed by conservative methods and require surgical intervention. The primary goals of surgical intervention are to relieve pain and mobilize the patient as soon as possible.

The aim of the study is to compare the short-term functional endoprosthetic recontruction, intramedullary nailing and open reduction internal fixation.

The primary tumor of the patient, applied chemotherapy and radiotherapy, Mirel risk score, Charlson comorbidity index, and PathFx 3.0 survival will be evaluated preoperatively.

The type of the operation will be decided at the multidisciplinary tumor council of ankara University.

ELIGIBILITY:
Inclusion Criteria:

* metastatic pathologic fracture
* operated via endoprosthesis, intramedullary nail or plate & screws

Exclusion Criteria:

* primary bone tumor
* conservative management
* neuromuscular disease
* periprosthetic fractures
* less than 1 month follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes patients with metastatic pathologic fractures treated via endoprosthesis, intramedullay nail or plate & screws.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal Tumor Society (MSTS) score | Preoperative
  MSTS score is for evaluating the patients with bone tumors. It consists of six domains; scored on a 0 to 5 scale and transformed into an overall score ranging from 0 to 100% with a higher score indicating better function.
Musculoskeletal Tumor Society (MSTS) score | Postoperative 1st day
  MSTS score is for evaluating the patients with bone tumors. It consists of six domains; scored on a 0 to 5 scale and transformed into an overall score ranging from 0 to 100% with a higher score indicating better function.
Musculoskeletal Tumor Society (MSTS) score | Postoperative 1st week
  MSTS score is for evaluating the patients with bone tumors. It consists of six domains; scored on a 0 to 5 scale and transformed into an overall score ranging from 0 to 100% with a higher score indicating better function.
Musculoskeletal Tumor Society (MSTS) score | Postoperative 1st month
  MSTS score is for evaluating the patients with bone tumors. It consists of six domains; scored on a 0 to 5 scale and transformed into an overall score ranging from 0 to 100% with a higher score indicating better function.
Toronto Extremity Salvage Score (TESS) | Preoperative
  TESS is widely used for the functional assessment of patients following surgery for musculoskeletal tumours. In the TESS system, specific movements for independent living and functionality are questioned and scored.While the worst score is 0, the best score for the lower extremity is 150, and the best score for the upper extremity is 145.
Toronto Extremity Salvage Score (TESS) | Postoperative 1st day
  TESS is widely used for the functional assessment of patients following surgery for musculoskeletal tumours. In the TESS system, specific movements for independent living and functionality are questioned and scored.While the worst score is 0, the best score for the lower extremity is 150, and the best score for the upper extremity is 145.
Toronto Extremity Salvage Score (TESS) | Postoperative 1st week
  TESS is widely used for the functional assessment of patients following surgery for musculoskeletal tumours. In the TESS system, specific movements for independent living and functionality are questioned and scored.While the worst score is 0, the best score for the lower extremity is 150, and the best score for the upper extremity is 145.
Toronto Extremity Salvage Score (TESS) | Postoperative 1st month
  TESS is widely used for the functional assessment of patients following surgery for musculoskeletal tumours. In the TESS system, specific movements for independent living and functionality are questioned and scored.While the worst score is 0, the best score for the lower extremity is 150, and the best score for the upper extremity is 145.
Visual analog scale (VAS) | Preoperative
  VAS is a widely used scale for pain. 0 means no pain where 10 means unbearable pain.
Visual analog scale (VAS) | Postoperative 1st day
  VAS is a widely used scale for pain. 0 means no pain where 10 means unbearable pain.
Visual analog scale (VAS) | Postoperative 1st week
  VAS is a widely used scale for pain. 0 means no pain where 10 means unbearable pain.
Visual analog scale (VAS) | Postoperative 1st month
  VAS is a widely used scale for pain. 0 means no pain where 10 means unbearable pain.
Upper Extremity Functional Scale (UEFS) | Preoperative
  UEFS is a functional scale for upper extremity. It is not specific for tumor patients.
Upper Extremity Functional Scale (UEFS) | Postoperative 1st day
  UEFS is a functional scale for upper extremity. It is not specific for tumor patients.
Upper Extremity Functional Scale (UEFS) | Postoperative 1st week
  UEFS is a functional scale for upper extremity. It is not specific for tumor patients.
Upper Extremity Functional Scale (UEFS) | Postoperative 1st month
  UEFS is a functional scale for upper extremity. It is not specific for tumor patients.
Disabilities of Arm, Shoulder and Hand (DASH) | Preoperative
  DASH is a widely used functional scale for upper extremity. It is not specific for tumor patients.
Disabilities of Arm, Shoulder and Hand (DASH) | Postoperative 1st day
  DASH is a widely used functional scale for upper extremity. It is not specific for tumor patients.
Disabilities of Arm, Shoulder and Hand (DASH) | Postoperative 1st week
  DASH is a widely used functional scale for upper extremity. It is not specific for tumor patients.
Disabilities of Arm, Shoulder and Hand (DASH) | Postoperative 1st month
  DASH is a widely used functional scale for upper extremity. It is not specific for tumor patients.
Lower Extremity Functional Scale (LEFS) | Preoperative
  LEFS is a functional scale for lower extremity. It is not specific for tumor patients.
Lower Extremity Functional Scale (LEFS) | Postoperative 1st day
  LEFS is a functional scale for lower extremity. It is not specific for tumor patients.
Lower Extremity Functional Scale (LEFS) | Postoperative 1st week
  LEFS is a functional scale for lower extremity. It is not specific for tumor patients.
Lower Extremity Functional Scale (LEFS) | Postoperative 1st month
  LEFS is a functional scale for lower extremity. It is not specific for tumor patients.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Preoperative
  WOMAC is a widely used functional scale for lower extremity. It is not specific for tumor patients.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Postoperative 1st day
  WOMAC is a widely used functional scale for lower extremity. It is not specific for tumor patients.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Postoperative 1st week
  WOMAC is a widely used functional scale for lower extremity. It is not specific for tumor patients.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Postoperative 1st month
  WOMAC is a widely used functional scale for lower extremity. It is not specific for tumor patients.

SECONDARY OUTCOMES:
Days at hospital after surgery | up to 1 month
  Hospitalization length required after the surgery.
Survival | up to 3 months
  Time that the patient lives after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty, Ankara, altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Final MSTS, TESS, UEFS, LEFS, DASH, WOMAC, VAS will be shared when the study is completed.